CLINICAL TRIAL: NCT03308851
Title: Evaluation of the Effects of Osteoperforation and Piezocorticision on Canine Retraction: Randomized Controlled Clinical Trial.
Brief Title: Evaluation of the Effects of Osteoperforation and Piezocorticision on Canine Retraction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulties related to COVID
Sponsor: Université de Montréal (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Le George Dinh-Khang, Principal investigator, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Piezo and Osteoperforation
Record Dates: First submitted 2017-10-02; First posted 2017-10-13 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Piezocorticision; Osteoperforation; Canine Retraction; Orthodontic Treatment

STUDY DESIGN:
Intervention Model Description: A split mouth design will be used where the experimental subjects will receive one procedure on one side of the upper dental arch and another procedure on the other side.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piezocorticision and osteoperforation group (Experimental): All participants in this arm will receive the piezocorticision and osteoperforation procedures on the upper jaw on the left and the right side.
  Interventions: Procedure: Piezocorticision; Procedure: Osteoperforation
- Control (No Intervention): The participants in this arm will receive no treatment, but will have the same monitoring as the experimental group.

INTERVENTIONS:
Procedure: Piezocorticision — The piezocorticision is a procedure that aims to accelerate the movement of teeth during an orthodontic treatment. It consists of a local anaesthesia followed by an incision of the buccal mucosa and an incision in the alveolar bone with a piezotome.
  Arms: Piezocorticision and osteoperforation group
Procedure: Osteoperforation — The osteoperforation is a procedure that aims to accelerate the movement of teeth during orthodontic treatment. It consists of a local anaesthesia followed by perforations of the buccal mucosa and alveolar bone using a specific osteoperforation tool.
  Arms: Piezocorticision and osteoperforation group

SUMMARY:
The primary objective of this research is to compare the rate of canine retraction following the osteoperforation and piezocorticision procedures in cases of first premolar extractions. The secondary objectives are to compare the second order movement of the canine (tipping), the amount of root resorption associated with the procedures, the inflammation process by measuring the inflammatory markers in the gingival crevicular fluid, the loss of posterior anchorage by measures on the cone beam computed tomography (CBCT) 3-dimensional radiograph and on the casts and to evaluate the pain level and the impact on quality of life following each procedure using the questionnaire of the visual analogue scale (VAS) of pain.

ELIGIBILITY:
Inclusion Criteria:

* Dental and/or skeletal Cl I and II requiring maxillary first premolar extraction.
* Young adults 16 years and older.
* Good overall health.
* Complete adult dentition.
* Cooperative.
* Acceptable hygiene.
* Absence of any periodontal disease (gingivitis, periodontitis).

Exclusion Criteria:

* Non-cooperative, fearful patients or patients with intellectual disability.
* Patients requiring the regular use of nonsteroidal anti-inflammatory drugs (NSAID).
* Use of antibiotics in the last 6 months.
* Previous or current use of bisphosphonates, corticosteroids or immunosuppressive drugs.
* Smokers.
* Patients suffering from uncontrolled systemic diseases (ex. diabetes type I and II).
* Presence of oral or maxillofacial malformations (ex. cleft palate) or dental pathologies (ex. ankylosis, abscess).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | From the time of force application until the distal of the canine touches the mesial of the second premolar. We estimate the time frame to be up to 24 weeks. Measures will be taken at two week intervals.
  The speed at which the canine is moved in the space of the extracted premolar.

SECONDARY OUTCOMES:
Amount of tipping | The measure is taken when the distal of the canine touches the mesial of the second premolar. We estimate the time frame to be up to 24 weeks
  The angulation of the long axis of the canine at the end of the retraction.
Amount of root resorption | The measure is taken when the distal of the canine touches the mesial of the second premolar. We estimate the time frame to be up to 24 weeks
  The total reduction in volume of the root of the canine caused by the canine retraction measured on the cone beam computed tomography.
Amount of posterior loss of anchorage | The measure is taken when the distal of the canine touches the mesial of the second premolar. We estimate the time frame to be up to 24 weeks
  Measure of the amount of anterior movement of the posterior teeth during the retraction of the canine.
Concentration of IL-1 in the gingival fluid sample | Measures are taken immediately before the periodontal procedures, then at 1,3,8 weeks and when the distal of the canine touches the mesial surface of the second premolar which can take up to 24 weeks.
  Measure of the concentration of IL-I using the Luminex technique.
Concentration of receptor activator of nuclear factor kappa-B ligand (RANKL) in the gingival fluid sample | Measures are taken immediately before the periodontal procedures, then at 1,3,8 weeks and when the distal of the canine touches the mesial surface of the second premolar which can take up to 24 weeks.
  Measure of the concentration of RANKL using the Luminex technique.
Concentration of osteoprotegerin (OPG) in the gingival fluid sample | Measures are taken immediately before the periodontal procedures, then at 1,3,8 weeks and when the distal of the canine touches the mesial surface of the second premolar which can take up to 24 weeks.
  Measure of the concentration of OPG using the Luminex technique.
Level of pain | Daily, for 7 days following extraction of premolars and piezocorticision and osteoperforation procedures
  Measure of the level of pain using a visual analogue scale of pain questionnaire ranging from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Clarice Nishio, D.M.D, MSc, PhD, Study Director — Université de Montréal
Locations (1):
- Clinique d'orthodontie de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03308851/Prot_000.pdf